CLINICAL TRIAL: NCT01702597
Title: The Effect of Whole Body Vibration and Acute Unilateral Unstable Lateral Ankle Sprain - A Biphasic Randomized Controlled Trial -
Brief Title: WBV and Acute Lateral Ankle Sprain
Acronym: WBV and ALAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Sebastian. F. Baumbach, Principle Investigator, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 315-12; MMW-Stiftung (Other: MMW-Stiftung)
Record Dates: First submitted 2012-10-03; First posted 2012-10-08 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Postural Control; Subjective Instablity
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- WBV (Experimental): Patients will receive supervised physical therapy using a whole body vibration device (Galileo® Med M Plus, Novotec, Pforzheim, Germany) twice a week, 30 minutes per session, for 6 weeks.
  Interventions: Device: Whole body vibration (Galileo® Med M Plus, Novotec, Pforzheim, Germany)
- Physiotherapy (Active Comparator): Patient will receive the current gold standard treatment protocol: supervised physical therapy, twice a week, 30 minutes per session, for 6 weeks.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Device: Whole body vibration (Galileo® Med M Plus, Novotec, Pforzheim, Germany) — Patients will train on a WBV platform, following a standardized protocol, aiming at improving strength, endurance and proprioception of both legs.
  Other Names: WBV; Galileo
  Arms: WBV
Other: Physiotherapy — Patients will receive a standardized physical therapy.
  Other Names: Physical Therapy, Training
  Arms: Physiotherapy

SUMMARY:
The aim of this bicentric, biphasic, randomized, controlled study is to compare of the current gold standard functional treatment to functional treatment plus WBV in patients with acute unilateral unstable inversion ankle sprains over a period of 12 months

DETAILED DESCRIPTION:
Background:

Ankle sprains often result in ankle instability, which is most likely caused by damage to passive and neurological structures. Whole body vibration (WBV) is a neuromuscular training method improving those neurologic parameters impaired. The aim of this study is to compare the current gold standard functional treatment to functional treatment plus WBV in patients with acute unilateral unstable inversion ankle sprains.

Methods/Design:

60 patients, aged 18-40 years, presenting with an isolated, unilateral, acute unstable inversion ankle sprain will be included in this bicentric, biphasic, randomized controlled trial. Patients will be randomized by envelope drawing. All patients will be allowed early mobilization and pain-depending weight bearing, limited functional immobilization by orthesis, PRICE, NSARDs as well as home and supervised physiotherapy. Supervised physical therapy will take place twice a week, 30 minutes per session, for 6 weeks, following a standardized intervention protocol. During supervised physical therapy, the intervention group will perform similar exercises on a side-alternating sinusoidal vibration platform as the control group. Two time dependent primary outcome parameters will be assessed. Short-term outcome after six weeks will be postural control quantified by the sway index. Mid-term outcome after one year will be assessed by subjective instability, defined by the presence of giving-way attacks. Secondary outcome parameters include return to pre-injury level of activities, residual pain, recurrence, objective instability, energy / coordination, Foot and Ankle Disability Index and EQ 5D.

ELIGIBILITY:
Inclusion Criteria:

* Acute, unilateral, unstable, inversion ankle sprain (Grade II, III)

Exclusion Criteria:

* Pregnancy
* Conditions affecting the neuromuscular- or musculoskeletal System
* Previous surgical interventions to the foot, ankle, knee or hip; known FAI, CAI
* Conditions possibly affecting balance
* Cardiovascular disease including thrombosis
* Respiratory diseases
* Abdominal diseases (including gallstones)
* Urological diseases (including kidney- and bladder stones)
* Gynaecological diseases and + intrauterine devices
* Neurological diseases including epilepsia within the last 2 years
* Acute injuries to the head
* Patient is not available for follow up visits
* Patient unable to give informed consent
* Patient suspected to be non-compliant

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Postural control | 6 weeks
  Sway Index measured via the Leonardo Mechanograph GRFP (16 bit, 800 Hz; NOVOTEC Medical GmbH, Germany)

SECONDARY OUTCOMES:
Subjective instability | 1 year
  Patient recorded giving-way symptoms or recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Schieker, Prof., Principal Investigator — Ludwig-Maximilians - University of Munich

REFERENCES:
- [Derived] Baumbach SF, Fasser M, Polzer H, Sieb M, Regauer M, Mutschler W, Schieker M, Blauth M. Study protocol: the effect of whole body vibration on acute unilateral unstable lateral ankle sprain- a biphasic randomized controlled trial. BMC Musculoskelet Disord. 2013 Jan 14;14:22. doi: 10.1186/1471-2474-14-22. PMID 23316791